CLINICAL TRIAL: NCT06721910
Title: Interplay Between Interleukin-6 and Glucagon in the Regulation of Human Amino Acid and Protein Homeostasis
Acronym: IGLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IGLU
Record Dates: First submitted 2024-03-30; First posted 2024-12-06 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Glucagon Resistance; Amino Acid Change
Keywords: interleukin-6; gluagon; pancreatic clamp
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Infusion of 100 ml normal saline
  Interventions: Other: Placebo
- IL-6R ab (Active Comparator): Infusion of tocilizumab, 8mg/kg body weight or max. 800mg in 100 ml normal saline
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Blockade of the interleukin-6 receptor
  Arms: IL-6R ab
Other: Placebo — Infusion of 100 ml normal saline
  Arms: Placebo

SUMMARY:
The goal of this proof-of-concept study is to learn if interleukin-6 changes the effect of glucagon in healthy volunteers. The main question it aims to answer is:

Does IL-6 influence how effectively glucagon lowers the concentration of amino acids in blood? Researchers will compare the infusion of normal saline and a blocker of the receptor for interleukin-6 to see if blocking interluekin-6 changes how effectively glucagon lowers the concentration of amino acids in blood.

Participants will be asked to

* receive either an infusion of normal saline or the interleukin-6 receptor blocker
* participate in a study visit three weeks later at which they will receive infusions of hormones and amino acids to mimic the concentrations of the hormones insulin and glucagon during fasting or fed conditions
* labelled glucose, glycerol and amino acids will also be infused continuously to track the fate of these molecules
* during the hormone infusions blood samples will be taken repeatedly

ELIGIBILITY:
Inclusion criteria:

* Age 18 to 50 years
* BMI 18.5 - 25 kg/m2
* Stable body weight in the past 6 months before study initiation
* Women should be anovulatory on non-cyclic hormone replacement or hormonal contraception

Exclusion criteria:

* Previous medical history for any chronic condition in the last three months, active disease or abnormal physical examination as verified by a qualified physician
* Body weight unstable in the past 6 months
* Use of tobacco/nicotine
* Alcohol consumption >30g/day
* Participation in an investigational drug trial within the past two months
* Current intake of any drugs (prescribed, over the counter or recreational)
* Known allergy to tocilizumab
* Pregnant or lactating women,
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Change in maximum glucagon-induced reduction in total plasma amino acid concentrations | At visit 2 during high glucagon phase (80-120 minutes)

SECONDARY OUTCOMES:
AUC of total amino acids | At visit 2 during high glucagon phase (80-120 minutes)
rate of phenylalanine oxidation | At visit 2 (15, 30, 45, 60, 80, 100, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300 minutes)
urea concentrations | At visit 2 (15, 30, 45, 60, 80, 100, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300 minutes)
rate of gluconeogenesis from amino acids | At visit 2 (15, 30, 45, 60, 80, 100, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300 minutes)
fractional synthesis rate of plasma proteins | At visit 2 (60, 180, 300 minutes)
Amino acid uptake by PBMCs ex vivo | At visit 1 and visit 2 (-120 minutes)
Change in fractional synthesis rate of lipoproteins | At visit 2 (60, 180, 300 minutes)
Cytokine plasma concentrations (IL-6, IL-1RA, TNF-alpha, IL-8, IL-10, CRP) | At visit 2 (15, 30, 45, 60, 80, 100, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300 minutes)
Plasma concentrations of insulin, c-peptide, glucagon, GH, IGF-1, cortisol, catecholamines, fT4, fT3, FGF21, follistatin, AGPTL4, ketones | At visit 2 (15, 30, 45, 60, 80, 100, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300 minutes)
Energy expenditure kcal/24 hours | At visit 2 (40, 160, 280 minutes)
Respiratory exchange rate | At visit 2 (40, 160, 280 minutes)
Oxygen consumption (VO2 ml/minutes) | At visit 2 (40, 160, 280 minutes)
Carbondioxid production (VCO2 ml/minutes) | At visit 2 (40, 160, 280 minutes)
Body composition (lean body mass kg) | At visit 1 and 2 (-120 minutes)
Body composition (fat bodymass kg) | At visit 1 and 2 (-120 minutes)
Blood pressure systolic | At visit 2 (-120 minutes)
Blood pressure diastolic | At visit 2 (-120 minutes)
Heart rate | At visit 2 (-120minutes)

OTHER OUTCOMES:
Changes in protein profiles | At visit 2 (60, 180, 300 minutes)
  Using untargeted and targeted proteomic platforms, the changes in protein profiles in the plasma will be measured
Changes in metabolite profiles | At visit 2 (60, 180, 300 minutes)
  Using untargeted and targeted metabolomic platforms, the changes in metabolite profiles in the plasma serum will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Beckey Trinh, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No